CLINICAL TRIAL: NCT04567602
Title: Non-Interventional Study on Pulmonary Arterial Hypertension Patients Treated With Macitentan or Selexipag: Experience From an Italian Cohort (INSPECTIO)
Brief Title: A Study of Pulmonary Arterial Hypertension Participants Treated With Macitentan or Selexipag
Acronym: INSPECTIO
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108855; 67896049PAH4009 (Other: Janssen-Cilag S.p.A., Italy)
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with PAH: Participants with confirmed diagnosis of pulmonary arterial hypertension (PAH) will be enrolled in the study and the data will be collected and observed to describe the application of European ESC/ERS guidelines and related 6th WSPH proceedings on risk assessment and related treatment strategy, in clinical practice.
  Interventions: Drug: PAH medication

INTERVENTIONS:
Drug: PAH medication — There will be no specific interventions.

SUMMARY:
The purpose of the study is to evaluate the change from baseline to 12 months after study enrollment in the number of the following non-invasive risk criteria: World Health Organization Functional Class (WHO/FC), 6-minute walk distance (6MWD), Brain Natriuretic Peptide (BNP) or N-terminal pro-brain Natriuretic Peptide (NT-proBNP).

ELIGIBILITY:
Inclusion Criteria:

* Participants in the clinical classification of pulmonary hypertension Group 1 (PAH)
* Participants with idiopathic, heritable and associated forms of PAH (connective tissue disease, congenital heart disease corrected at least 1-year ago, human immunodeficiency virus infection, drug use or toxin, and porto-pulmonary)
* Confirmed diagnosis of PAH with hemodynamic study right heart catheterization (RHC) at enrolment or at latest follow-up (not later than twelve months from enrolment date)
* Participants with a low or intermediate mortality risk profile, as per clinical judgement based on a multiparametric approach including clinical, functional exercise, right ventricular function and hemodynamic parameters
* Participants currently in treatment with selexipag and/or macitentan (in monotherapy or in combination therapy)

Exclusion Criteria:

* Participants in Group 1 that are responders to the vasoreactivity test
* Participants with pulmonary veno-occlusive disease (PVOD), defined on the basis of the following chest findings at high-resolution computed tomography (HRCT): centrilobular ground-glass opacities, smooth thickening of interlobular septa, mediastinal lymph node enlargement
* Participants already in treatment with subcutaneous/intravenous prostanoids. Iloprost interventional (IV) (treatment of digital ulcers in systemic sclerosis [SSc] participants according to european league against rheumatism [EULAR] guidelines) is allowed
* Participants currently enrolled in an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consist of participants with confirmed diagnosis of PAH.
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Number of the Non-Invasive Low-Risk Criteria to 12 Months | Baseline and 12 Months
  Change from baseline in the number of the non-invasive low-risk criteria will be assessed according to the following parameters: world health organization (WHO)/functional class (FC)- I, II, 6-minute walk distance (6MWD) greater than (>) 440 meters (m), and brain natriuretic peptide (BNP) less than (<) 50 nanogram per liter (ng/l) or N-terminal-pro-hormone brain natriuretic Peptide (NT-proBNP) <300 ng/l.

SECONDARY OUTCOMES:
Number of Participants with Improved, Stable or Worsened Risk profile from Baseline to 12 and 24 Months | Baseline up to 12 and 24 Months
  Risk profile is assessed as improved, stable or worsened where improved indicates 1 or more non-invasive parameters from intermediate to low risk profile; stable indicates no change in the parameters; and worsened indicates 1 or more non-invasive parameters move from low or intermediate to intermediate or high range risk.
Change in Progression in the Number of Participants with Low/High Intermediate Risk | Baseline up to 24 Months
  Change in risk profile for the low/high intermediate risk participants according to following cut-off values for low intermediate risk/high intermediate risk, respectively: (6MWD [greater than or equal to [>=] or < 300m], Peak oxygen consumption [VO2] [>= or < 50% predicted], BNP [less than or equal to [<=] or > 175 ng/l], or NT-proBNP [<= or > 850 ng/l], right atrial area [RA] [<= or > 22 centimeter [cm]] and right atrial pressure [RAP] [<= or > 11 millimeter of mercury [mmHg]] or stroke volume index (SVI) (> or <= 38 milliliter per meter square [ml/m2])). The low intermediate risk is defined by a presence of at least three low intermediate parameters and a high intermediate risk is defined by a presence of at least three high intermediate parameters.
Change from Baseline in 6MWD | Baseline up to 24 Months
  Change from baseline in 6MWD will be reported.
Change from Baseline in BNP or NT-proBNP | Baseline up to 24 Months
  Change from baseline in BNP or NT-proBNP will be reported.
Change from Baseline in Registry to Evaluate Early and Long-term PAH Disease Management (REVEAL) 2.0 Risk Score up to 12 and 24 Months | Baseline up to 12 and 24 Months
  The REVEAL risk calculator determines the risk status and the scores can be defined as: low risk as a score of <= 6, intermediate risk as a score of 7 or 8, and high risk as a score of >= 9 for the survival rates.
Adherence to European Society of Cardiology and European Respiratory Society (ESC/ERS) guidelines and 6th World Symposium on Pulmonary Hypertension (WSPH) | Up to 24 Months
  Adherence to ESC/ERS guidelines and 6th WSPH will be reported.
Change from Baseline in Echocardiographic Parameters | Baseline up to 24 Months
  Change in echocardiographic parameters will be reported as assessed by echocardiogram.
Change from Baseline in Hemodynamic Parameters | Baseline up to 24 Months
  Change in hemodynamic parameters will be reported.
Hospitalization Rate due to Worsening of PAH | Up to 24 Months
  The hospitalization rate due to PAH worsening will be calculated based on the number of participants with at least one hospitalization. The calculation of the rate will be based on the number of events over the whole follow-up time that is exposure time.
Overall Survival (OS) | Up to 24 Months
  OS is defined as the duration/time from the start of study treatment to date of death due to any cause.
Change from Baseline in Health-Related Quality of Life (HRQoL) as Measured with Emphasis-10 Questionnaire | Baseline up to 24 Months
  The emPHasis-10 is a short and easy questionnaire that consists of 10 items which address breathlessness, fatigue, control and confidence. Each item is scored on a semantic differential six-point scale (0-5), with contrasting adjectives at each end. A total emPHasis-10 score is derived using simple aggregation of the 10 items. emPHasis-10 scores range from 0 to 50, higher scores indicate worse quality of life.
Change from Baseline in Participants with Narrative plots | Baseline and 12 Months
  Participants will be invited to fill in two narrative plots; one at the enrollment visit and one at the month 12 visit.
Change from Baseline in Caregivers with Narrative Plots | Baseline and 12 Months
  Caregivers will be invited to fill in two narrative plots; one at the enrollment visit and one at the month 12 visit.
Number of Participants with Adverse Events (AEs) and Adverse Drug Reactions (ADRs) | Up to 24 Months
  An AE is any untoward medical occurrence in a participant enrolled in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. An ADR is defined as a response to a medicinal (investigational or non-investigational) product that is noxious and unintended.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.p.A., Italy Clinical Trial, Study Director — Janssen-Cilag S.p.A.
Locations (30):
- Italy (30):
  - Generale Regionale F. Miulli, Acquaviva delle Fonti
  - A.O. Universitaria Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - Ospedale Di Venere, Bari
  - Ospedale di Bolzano, Bolzano
  - ASST Spedali Civili Brescia, Brescia
  - Azienda Ospedaliera G. Brotzu, Cagliari
  - AO di Catanzaro Pugliese Ciaccio, Catanzaro
  - ASL2 Lanciano - Vasto - Chieti - Ospedale 'SS Annunziata' di Chieti, Chieti
  - AOU Careggi, Florence
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Foggia, Foggia
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Presidio Ospedaliero di Ivrea, Ivrea
  - UOC Oncologia Ospedale Provinciale di Macerata, Macerata
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Centro Cardiologico Monzino, Milan
  - Ospedale Monaldi, Napoli
  - Università del Piemonte Orientale - Ospedale Maggiore della Carità di Novara, Novara
  - AOU di Padova, Padua
  - ISMETT Istituto Mediterraneo Trapianti e Terapie ad Alta Specializzazione, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Toscana Gabriele Monasterio CNR, Pisa
  - AOU Policlinico Umberto I, Roma
  - Policinico A Gemelli, Roma
  - IRCCS Policlinico San Donato, San Donato Milanese
  - Presidio SS Annunziata AOU Sassari, Sassari
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
  - ASUI Santa Maria della Misericordia di Udine, Udine
  - Ospedale Borgo Roma, Verona